CLINICAL TRIAL: NCT02286180
Title: Job Stress and Frontal Activity During Verbal Fluency Test: A Near-infrared Spectroscopy Study
Brief Title: Subjective Feelings of Job Stress and Frontal Activity During Verbal Fluency Test: A Near-infrared Spectroscopy Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, TCVGH, Attending Physician, Taichung Veterans General Hospital
Other Study IDs: CF14045
Record Dates: First submitted 2014-11-04; First posted 2014-11-07 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Stress
Keywords: near infrared spectroscopy; NIRS; intern

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
Background and objectives:

Recently the news of intern doctors' death due to overloaded work or committing suicide has made the authorities concerned put emphasis on the mental health care of medical staffs and related policies of psychological interventions. The prefrontal lobe plays an important role in the working memory, executive function and problem-solving abilities of the brain. Currently, no neuroimaging studies investigating the impact of job stress on the prefrontal love functions in intern doctors. Functional near-infrared spectroscopy (fNIRS) measures the cortical functions of the frontotemporal regions and has been widely used as a biomarker to aid in differential diagnoses in major psychiatric illnesses in Japan. The present study will investigate impact of the job stress on brain cortical activity during a verbal fluency test (VFT) by using fNIRS.

Materials and methods:

A total of 100 participants will be recruited. Clinical measurements of mood status by Beck's Depression Inventory and Beck's Anxiety Inventory, as well as job stress by Chinese Version of the Job Content Questionnaire and the Chinese version of Copenhagen Burnout Inventory will be arranged. The relationship between clinical measurements and cortical activity during a VFT will be analyzed by Pearson's correlation. Multiple regression analysis will be applied to investigate the independent contributions of mood status and job stress.

Expected results and contributions of the study:

Job stress, depression, and anxiety are significantly negatively correlated with cortical activity of prefrontal regions. The importance of mental health of medical staffs under high job stress should be stressed.

DETAILED DESCRIPTION:
A total of 100 intern doctors will be recruited. The data including Chinese version of Copenhagen burnout inventory, BDI, BAI, average working hours per day, and average sleeping times were acquired. They will undergo NIRS investigations to detect frontal activities during performing a verbal fluency test. The correlation between stress parameters and cortical activities were examined.

ELIGIBILITY:
Inclusion Criteria:

* medical intern doctors who are willing to participate in the study.

Exclusion Criteria:

* with past psychiatric disease
* with history substance abuse or dependence
* with history neurological disorders or head trauma

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medical Intern Doctors in a medical center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
frontal cortical activities during cognitive test detecting by near infrared spectroscopy | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: PoHan Chou, MD, Principal Investigator — Taichung Veterans General Hospital, Taiwan, ROC.